CLINICAL TRIAL: NCT06054126
Title: The Development of Coronary Collateralization in Type 2 Diabetic Patients With Chronic Total Occlusion
Brief Title: COronary CoLLateralization in Type 2 diabEtic Patients With Chronic Total Occlusion
Acronym: COLLECT
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: sy11218
Record Dates: First submitted 2023-09-19; First posted 2023-09-26 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-08

CONDITIONS: Chronic Total Occlusion of Coronary Artery; Diabetes Mellitus, Type 2
Keywords: Atherosclerosis; Diabetes Mellitus, Type 2; Chronic Total Occlusion of Coronary Artery; Coronary artery disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Atherosclerosis; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — plasma and PBMCs
Oversight: FDA-regulated Device: No

GROUPS / COHORTS (2):
- T2DM with good CCC: T2DM was diagnosed according to the criteria of the American Diabetes Association. The diagnosis of CTO was made if at least one lesion was angiographic 100% occlusion. Coronary collateral circulation development was graded according to the Cohen-Rentrop method, grade 2 (partial filling of the epicardial segment by collateral vessels); grade 3 (complete filling of the epicardial artery by collateral vessels) were defined as good coronary collateral circulation.
  Interventions: Other: Echocardiography
- T2DM with poor CCC: T2DM was diagnosed according to the criteria of the American Diabetes Association. The diagnosis of CTO was made if at least one lesion was angiographic 100% occlusion. Coronary collateral circulation development was graded according to the Cohen-Rentrop method, grade 0 (no filling of any collateral vessels) and grade 1 (filling of side branches of the artery to be perfused by collateral vessels without visualization of the epicardial segment) were defined as poor coronary collateral circulation.
  Interventions: Other: Echocardiography

INTERVENTIONS:
Other: Echocardiography — Cardiac function was evaluated by echocardiography at one year follow-up.

SUMMARY:
A severe coronary artery obstruction is a prerequisite for spontaneous collateral recruitment. The formation of coronary collateral circulation(CCC) is significantly impaired in type 2 diabetic patients with chronic total occlusion (CTO) compared with non-diabetic patients with CTO. This retrospective cohort enrolls consecutive T2DM patients who had at least one lesion with coronary angiographic total occlusion.

DETAILED DESCRIPTION:
COronary CoLLateralization in Type 2 diabEtic Patients With Chronic Total Occlusion (COLLECT) study is a single center, retrospective cohort study to investigate potential factors associated with the development of coronary collateral circulation in diabetic patients. Investigators will consecutively enroll T2DM patients who had at least one lesion with coronary angiographic total occlusion. The development of coronary collateral circulation will be graded according to the Rentrop method and patients will be divided into poor CCC (grade 0 or 1) or good (grade 2 or 3) CCC groups according to their Rentrop grades. Baseline clinical and laboratory characteristics at hospital admission will be recorded to analyze potential factors associated with the development of coronary collateral circulation in T2DM patients with CTO. Later, their cardiac function will be evaluated by echocardiography at one year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-90 years
* Type 2 diabetes diagnosed by one of the following criteria:

HbA1c >/= 6.5% Fasting plasma glucose >/= 7.0 mmol/l (confirmed) 2h plasma glucose value during OGTT >/= 11.1 mmol/l Already receiving glucose-lowering agents.

* At least one lesion with angiographic total occlusion

Exclusion Criteria:

* eGFR<15mL/(min·1.73m2)
* chronic heart failure with NYHA grade ≥3
* had a history of coronary artery bypass grafting
* had received a percutaneous coronary intervention within the prior 3 months
* Malignant tumor or immune system disorders
* Pulmonary heart disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetic patients with chronic total occlusion undergone coronary angiography at Ruijin Hospital, Shanghai, China are consecutively enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Cardiac function evaluated by echocardiography | 12 months
  Assessed by echocardiography

SECONDARY OUTCOMES:
Cardiovascular events | up to 5 years
  The incidence of MACCE (major adverse cardiac and cerebrovascular events)

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mao LS, Wang YX, Qi Y, Yue ZR, Ding FH, Wang XQ, Lu L, Shen WF, Shen Y. Elevated Uric Acid/Albumin Ratio Predicts Poor Coronary Collateral Circulation in Type 2 Diabetic Patients With Stable Coronary Artery Disease. J Diabetes Res. 2025 Dec 19;2025:9721061. doi: 10.1155/jdr/9721061. eCollection 2025. PMID 41497488
- [Derived] Mao LS, Geng L, Wang YX, Qi Y, Wang MH, Ding FH, Dai Y, Lu L, Zhang Q, Shen WF, Shen Y. Clinical risk score to predict poor coronary collateralization in type 2 diabetic patients with chronic total occlusion. BMC Cardiovasc Disord. 2025 Apr 2;25(1):250. doi: 10.1186/s12872-025-04687-8. PMID 40175898